CLINICAL TRIAL: NCT07394322
Title: The Role of Serum of Interleukin-6 in Predicting the Development of Meconium Aspiration Syndrome in Infants Born With Meconium-Stained Amniotic Fluid
Brief Title: Interleukin-6 in the Development of Meconium Aspiration Syndrome in Newborn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Nashwa farouk Mohamed, lecturer of pediatrics, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MS-15-1-2022
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Meconium Aspiration Syndrome
Keywords: Meconium aspiration syndrome IL-6: interleukin-6
MeSH Terms: conditions — Meconium Aspiration Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 120 term newborns who were born from mothers who had MSAF & admitted to NICU at Benha University hos (Experimental): 120 term newborns who were born from mothers who had MSAF & admitted to NICU at Benha University hospitals for a period of 1year, starting from February 2022 to February 2023 (Approval No: MS-15-1-2022). Patients were divided according to outcome into two groups: Group 1 (MAS group) contained 60 neonates who developed meconium aspiration syndrome, & Group 2 (control group) involved 60 neonates who did not develop meconium aspiration syndrome.
  Interventions: Diagnostic Test: serum interleukin 6

INTERVENTIONS:
Diagnostic Test: serum interleukin 6 — Serum IL-6: An enzyme-linked immunosorbent test (ELISA) that was developed to quantify the amount of the target bound amongst a matched pair of antibodies was the Human IL-6 solid-phase sandwich ELISA. The wells of the microplate that were provided already had a target-specific antibody coated on them. After that, the immobilized (captured) antibody was bound to samples, standards, or controls by adding them to these wells. Using the second antibody to make a sandwich with the enzyme, antibody, and target complex, a substrate solution was added to make a signal that could be picked up. This signal's strength was proportionate to the original specimen's target concentration.
  Steps: To achieve the desired result, remove the desired number of strips & allow them to reach room temperature. Two to eight degrees Celsius was the temperature at which the unused strips as well as the desiccant were placed back into the sealed aluminum foil bag. The blank wells should be set aside (if the measur

SUMMARY:
This trial is intended to assess the serum levels of interleukin-6 as a predictive factor for the occurrence of meconium aspiration syndrome in infants born with MSAF.

DETAILED DESCRIPTION:
Meconium aspiration syndrome happens when a baby inhales a combination of meconium (the first stool) as well as amniotic fluid into their lungs during the delivery process. Meconium aspiration syndrome is a prevalent reason for significant respiratory failure in full-term or post-term newborns. MAS fluid is responsible for around 8 to 19% of all term deliveries, and meconium aspiration syndrome develops in around five to thirty-three percent of these infants (1).

Interleukin-6 is classified as a cytokine. One of the mediators of inflammation released early in septic shock is critical for initiating the immune response. It also has a role in activating T lymphocytes and B lymphocytes, as well as encouraging lymphocyte proliferation and differentiation. Furthermore, IL-6 possesses strong pyrogenic properties. Additionally, it stimulates the secretion of acute-phase proteins like CRP (2).

IL-6 is a powerful inflammatory agent, as well as its level in the blood has been assessed as a predictive marker in many studies. It is considered one of the foremost indications of prenatal inflammation. Raised levels of interleukin-6 are also observed in both infectious & non-infectious inflammatory and stressful conditions (2, 3).

Nonspecific symptoms such as a rise in breathing in flattening of the diaphragm, radiography & irregular linear or patchy patches of atelectasis are observed during the early phase of meconium aspiration syndrome. These signs are present in the early stages of syndrome. However, characteristic indications, for instance, extensive, coarse, and evenly distributed opacities resulting from pneumonia & interstitial edema, may not manifest until 2-3 days later. Therefore, it is necessary to use indicators to predict whether people are prone to developing MAS. The role of inflammation in the progression of MAS is acknowledged (4).

Prior studies have shown that cytokine levels in Meconium aspiration syndrome experience an elevation in both controlled laboratory conditions (in vitro) as well as living creatures (in vivo) (5).

ELIGIBILITY:
Inclusion Criteria:

* both genders (Males and females), term infants (above 37 gestational weeks), and born from ladies who have meconium-stained amniotic fluid.

Exclusion Criteria:

* Infants born to mothers suspected of having chorioamnionitis (leukocytosis, fever, early membrane rupture (above 18 hours), foul-smelling discharge, tachycardia in the mother or fetus, as well as a positive blood culture),
* those without parental consent,
* those with severe perinatal asphyxia (Stage two or three of hypoxic-ischemic encephalopathy findings according to Sarnat (6)),
* those with severe chorioamnionitis,
* those withcongenital abdominal malformations,

Ages: 1 Minute to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
serum IL-6 | in 3 days of delivery
  Serum IL-6: An enzyme-linked immunosorbent test (ELISA) that was developed to quantify the amount of the target bound amongst a matched pair of antibodies was the Human IL-6 solid-phase sandwich ELISA
: Evaluating the levels of interleukin-6 (IL-6) in the blood serum to determine its ability to predict the occurrence of MAS in newborns delivered with meconium-stained amniotic fluid. | in 3 days of delivery
  Serum IL-6: An enzyme-linked immunosorbent test (ELISA) that was developed to quantify the amount of the target bound amongst a matched pair of antibodies was the Human IL-6 solid-phase sandwich ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Benha Faculty of Medicine, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: No